CLINICAL TRIAL: NCT01706263
Title: U0289-402: An Open Label, 8 Week Study to Evaluate the Efficacy and Tolerability of MAXCLARITY II in Subjects With Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114551
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Salicylic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MAXCLARITY II (Experimental): MAXCLARITY II (2.5% BPO) Foam Cleanser and Foam Treatment and (0.5% Salicylic Acid) Toner Foam. Available over-the-counter.
  Interventions: Drug: MAXCLARITY II (2.5% BPO) Foam Cleanser; Drug: MAXCLARITY II (2.5% BPO) Foam Treatment; Drug: MAXCLARITY II (0.5% Salicylic Acid) Toner Foam

INTERVENTIONS:
Drug: MAXCLARITY II (2.5% BPO) Foam Cleanser — Available over the counter.
Drug: MAXCLARITY II (2.5% BPO) Foam Treatment — Available over the counter.
Drug: MAXCLARITY II (0.5% Salicylic Acid) Toner Foam — Available over the counter.

SUMMARY:
One of the main success factors in acne therapy is user compliance with treatment, product cost, availability and ease of use. Poor compliance may translate into decreased efficacy (either not improving symptoms well enough or not improving symptoms fast enough), tolerability issues or adverse effects (eg, erythema, dryness, or peeling of the skin), a lack of understanding of the instructions for use, or product cost/availability. Whatever the reason, poor compliance translates to decreased efficacy and increased frustration on the part of the user.

The current study will evaluate the efficacy and tolerability of MAXCLARITY II, an over the counter, topical benzoyl peroxide (BPO) product line, in subjects with acne.

DETAILED DESCRIPTION:
Acne vulgaris is an extremely common dermatological disease that is found typically in adolescence and young adulthood. Acne vulgaris manifests with open and closed comedones (blackheads and whiteheads), papules, pustules, nodules, and cysts on the face, neck, and trunk. Scarring can occur, particularly if the lesions are inflamed and deep, even in the absence of external manipulation (eg, picking and squeezing) of the skin.

Acne vulgaris can be treated with a variety of agents that are selected to address the pathogenic factors assumed to be responsible for the type and degree of manifested acne lesions. Monotherapy and combination therapy regimens are both useful. Topical agents are generally used as first-line therapy and include retinoids, antibiotic preparations (eg, erythromycin and clindamycin), benzoyl peroxide (BPO), alpha and beta hydroxy acids (eg, glycolic and salicylic acid preparations), and azelaic acid. Systemic therapies are initiated in patients with moderate to severe inflammatory acne that does not respond to topical therapy.

Benzoyl peroxide has antimicrobial and anti inflammatory properties and is often considered an important component of acne treatment. Benzoyl peroxide is frequently the first product that adolescents will use for acne because it can be purchased without a prescription in several different concentrations and formulations.

One of the main success factors in acne therapy is user compliance with treatment, product cost, availability and ease of use. Poor compliance may translate into decreased efficacy (either not improving symptoms well enough or not improving symptoms fast enough), tolerability issues or adverse effects (eg, erythema, dryness, or peeling of the skin), a lack of understanding of the instructions for use, or product cost/availability. Whatever the reason, poor compliance translates to decreased efficacy and increased frustration on the part of the user.

The current study will evaluate the efficacy and tolerability of MAXCLARITY II, an over the counter, topical benzoyl peroxide (BPO) product line, in subjects with acne.

This is a multi center, open label study to evaluate the efficacy and tolerability of MAXCLARITY II, an over the-counter, topical benzoyl peroxide product line, in subjects with acne. Approximately 30 subjects, aged from 16 to 29 years, inclusive, with mild facial acne vulgaris are expected to participate in the study. No more than 50% of the subjects at each site can be enrolled under the age of 20.

An expert grader will complete counts of inflamed lesions (papules/pustules) and noninflamed lesions (open/closed comedones), the ISGA, and an assessment of tolerability at each study visit. Subjects will assess tolerability at each study visit and will complete a product acceptability and preference questionnaire at the end of the study.

The study duration will be 8 weeks (56 days) with visits at baseline (day 1), week 1, week 2, week 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
2. Male or female aged from 16 to 29 years, inclusive, at time of consent. No more than 50% of the subjects at each site can be enrolled under the age of 20.
3. Mild facial acne vulgaris, characterized by at least 24 facial inflammatory lesions (papules and pustules) and/or noninflammatory lesions (open and closed comedones) on the face.
4. Able to complete the study and to comply with study instructions.
5. Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Acceptable contraceptive methods include the following:

   * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of nonhormonal contraception should be added until the third continuous month of hormonal contraception has been completed.
   * Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided that the female subject has never given birth naturally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal sterilization or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermatocide is acceptable.
   * Women who are not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the study.

Exclusion Criteria:

1. Female who is pregnant, trying to become pregnant, or breast feeding.
2. Has active or chronic skin allergies.
3. Has a history of acute or chronic disease that might interfere with or increase the risk of study participation.
4. Had skin cancer treatment in preceding 12 months.
5. Has damaged skin on facial areas (eg, sunburn, tattoo, or scar)
6. Had any medical procedure (eg, laser resurfacing, chemical peel, or plastic surgery) on facial areas in preceding 12 months.
7. Had any cosmetic procedure (eg, microdermabrasion) on facial areas within 8 weeks of the baseline visit.
8. Has any dermatological disorder that in the opinion of the investigator may interfere with the accurate evaluation of the subject's facial appearance.
9. Received any investigational drug or procedure within 28 days of the baseline visit or is scheduled to receive an investigational drug (other than the study products) or procedure during the study.
10. Currently using any medication that in the opinion of the investigator may affect the evaluation of the study products or place the subject at undue risk (including but not limited to asthma medications, oral steroids, rifampin, anticonvulsants, and St John's wart).
11. Has a history of known or suspected intolerance to any of the ingredients of the study products (ie, benzoyl peroxide).
12. Considered unable or unlikely to attend the necessary visits.
13. Live in the same household as currently enrolled subjects.
14. Employee of the investigator, a contract research organization, or Stiefel Laboratories who is involved in the study, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2009-11-20 (Actual); Study Completion 2009-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114551 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114551 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114551 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114551 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114551 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114551 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female participants aged from 18 to 29 years with mild facial acne vulgaris were enrolled in this study. The study was conducted at three different study centers. Study period was 8 Weeks (56 days) and study conducted from 19 August 2009 to 01 December 2009.
Groups:
- MAXCLARITY II: The eligible participants applied a small amount of the MAXCLARITY II™ 2.5 percent (%) benzyl peroxide foam cleanser and foam treatment, 0.5% salicylic acid toner foam. Participants applied foam cleanser each morning to the dampened skin and gently massaged over whole face followed by thorough wash with warm water. The participants then applied small amount of MAXCLARITY II foam treatment in a thin layer to the entire face (avoiding the eyes, lips, and mouth) each morning. In the evening the participants washed their face with MAXCLARITY II Foam cleanser and then applied MAXCLARITY II toner foam to the face each evening. Study products were applied once daily for 8 weeks. If any dose was missed, the next dose was administered according to original schedule.
Period: Overall Study
Arm/Group | MAXCLARITY II
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MAXCLARITY II: The eligible participants applied a small amount of the MAXCLARITY II 2.5 % benzyl peroxide foam cleanser and foam treatment, 0.5% salicylic acid toner foam. Participants applied foam cleanser each morning to the dampened skin and gently massaged over whole face followed by thorough wash with warm water. The participants then applied small amount of MAXCLARITY II foam treatment in a thin layer to the entire face (avoiding the eyes, lips, and mouth) each morning. In the evening the participants washed their face with MAXCLARITY II Foam cleanser and then applied MAXCLARITY II toner foam to the face each evening. Study products were applied once daily for 8 weeks. If any dose was missed, the next dose was administered according to original schedule.
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Inflammatory, Non Inflammatory, and Total Lesion Counts From Baseline to Week 8
Description: Evaluator assessed the left and right side of the face as inflammatory (papules [solid elevation of skin with no visible fluid] and pustules [small inflamed elevation of the skin that is filled with pus]) and non-inflammatory (open [blackheads] and closed [whiteheads] comedones) and total lesions (sum of inflammatory and non-inflammatory lesion) for each participant. Each type of lesion was counted separately; the lesion counts were taken from the face from hairline to the mandible (including forehead, cheeks, and chin). Total lesion counts were calculated as the sum of the inflammatory and non-inflammatory lesion counts. Percent change from Baseline to Week 8 was calculated as the value at Week 8 minus the value at Baseline divided by the Baseline value multiplied by 100. Baseline was defined as Day 1 value .
Time Frame: Baseline (Day 1) and Week 8
Population: Intent-to-treat analysis set was used which included data from all randomized participants who received study product.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Percent change
  Inflammatory lesion count | -62.1 (37.1)
  Non-Inflammatory lesion count | -49.8 (39.7)
  Total lesion count | -56.9 (32.7)

2. Secondary Outcome: Mean Percent Change in Inflammatory, Non Inflammatory, and Total Lesion Counts From Baseline to Weeks 1, 2, and 4
Description: Evaluator assessed the left side and right side of the face as inflammatory (papules [solid elevation of skin with no visible fluid] and pustules [small inflamed elevation of the skin that is filled with pus]) and non-inflammatory (open comedones [blackheads] and closed comedones [whiteheads]) and total lesions for each participant. Each type of lesion was counted separately; the lesion counts were taken from the face from hairline to the mandible (including forehead, cheeks, and chin). Total lesion counts was calculated as the sum of the inflammatory and non-inflammatory lesion counts. Percent change from Baseline to specified time (Weeks 1, 2, and 4) point was calculated as the value at specified time point minus the value at Baseline divided by the Baseline value multiplied by 100. Baseline was defined as Day 1 value .
Time Frame: Baseline (Day 1) and Week 1, 2, 4
Population: Intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Percent change
  Inflammatory lesion count, Week 1 | -27.9 (29.8)
  Inflammatory lesion count, Week 2 | -50.8 (25.6)
  Inflammatory lesion count, Week 4 | -49.5 (30.6)
  Non-Inflammatory lesion count, Week 1 | -9.9 (45.1)
  Non-Inflammatory lesion count, Week 2 | -23.4 (38.0)
  Non-Inflammatory lesion count, Week 4 | -34.3 (37.5)
  Total lesion count, Week 1 | -22.6 (27.6)
  Total lesion count, Week 2 | -37.8 (24.1)
  Total lesion count, Week 4 | -44.9 (28.5)

3. Secondary Outcome: Mean Change in Investigator's Static Global Assessment (ISGA) From Baseline to Weeks 1, 2, 4 and 8
Description: Evaluator assessed the acne severity of participants' faces using the ISGA scale on a five point scale which ranged from 0 to 4 defined as 0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe. Change from Baseline to specified time point (Weeks 1, 2, 4 and 8) was calculated as the value at specified time point minus the value at Baseline. Baseline was defined as Day 1 value .
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8
Population: Intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Score on a scale
  ISGA score, Week 1 | -0.07 (0.54)
  ISGA score, Week 2 | -0.46 (0.58)
  ISGA score, Week 4 | -0.39 (0.69)
  ISGA score, Week 8 | -0.61 (0.69)

4. Secondary Outcome: Percentage of Participants Who Improved by at Least One Grade on the ISGA
Description: Evaluator assessed the acne severity of participants' faces using the ISGA scale on a five point scale which ranged from 0 to 4 defined as 0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe. Percent change from Baseline to specified time point was calculated as the value at specified time point minus the value at Baseline divided by the Baseline value multiplied by 100. Baseline was defined as Day 1 value .
Time Frame: Up to Week 8
Population: Intent-to-treat analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Percentage of participants
  Atleast one grade improvement,Week 1 | 17.9
  Atleast two grade improvement,Week 1 | 0.0
  Atleast one grade improvement,Week 2 | 42.9
  Atleast two grade improvement,Week 2 | 3.6
  Atleast one grade improvement,Week 4 | 35.7
  Atleast two grade improvement,Week 4 | 7.1
  Atleast one grade improvement,Week 8 | 50.0
  Atleast two grade improvement,Week 8 | 10.7

5. Secondary Outcome: Change in Investigator Assessment of Tolerability (Erythema, Dryness and Peeling) From Baseline to Weeks 1, 2, 4 and 8.
Description: Erythema , dryness, and peeling, were evaluated independently by the investigator on a five point scale ranged from 0 to 4 defined as 0-none, 1-very minimal, 2-mild, 3-moderate, 4-severe. Change from Baseline to specified time point (Weeks 1, 2, 4 and 8) was calculated as the value at specified time point minus the value at Baseline. Baseline was defined as Day 1 value .
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8
Population: Intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Score on scale
  Erythema, Week 1 | 0.00 (0.38)
  Erythema, Week 2 | -0.04 (0.43)
  Erythema, Week 4 | -0.04 (0.79)
  Erythema, Week 8 | -0.32 (0.55)
  Dryness, Week 1 | 0.14 (0.45)
  Dryness, Week 2 | 0.32 (0.61)
  Dryness, Week 4 | 0.11 (0.42)
  Dryness, Week 8 | 0.11 (0.31)
  Peeling, Week 1 | 0.11 (0.42)
  Peeling, Week 2 | 0.21 (0.50)
  Peeling, Week 4 | 0.04 (0.19)
  Peeling, Week 8 | 0.11 (0.31)

6. Secondary Outcome: Change in Participant Assessment of Tolerability (Redness, Dryness, Burning, Itching and Scaling) From Baseline to Weeks 1, 2, 4 and 8
Description: Redness, dryness, burning, itching and scaling were evaluated independently by the participant on a five point scale ranged from 0 to 4 defined as 0-none, 1-very minimal, 2-mild, 3-moderate, 4-severe. Change from Baseline to specified time point (Weeks 1, 2, 4 and 8) was calculated as the value at specified time point minus the value at Baseline. Baseline was defined as Day 1 value .
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8
Population: Intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MAXCLARITY II
Number analyzed (Participants) | 28
Score on scale
  Redness,Week 1 | -0.39 (1.03)
  Redness,Week 2 | -0.25 (1.24)
  Redness,Week 4 | -0.18 (1.09)
  Redness,Week 8 | -0.36 (1.34)
  Dryness,Week 1 | 0.04 (1.20)
  Dryness,Week 2 | 0.07 (1.30)
  Dryness,Week 4 | 0.00 (1.09)
  Dryness,Week 8 | 0.11 (1.40)
  Burning,Week 1 | 0.21 (1.10)
  Burning,Week 2 | 0.36 (1.22)
  Burning,Week 4 | 0.32 (0.67)
  Burning,Week 8 | -0.07 (1.02)
  Itching,Week 1 | 0.07 (0.90)
  Itching,Week 2 | 0.07 (1.02)
  Itching,Week 4 | 0.14 (1.15)
  Itching,Week 8 | 0.07 (0.94)
  Scaling,Week 1 | -0.14 (0.71)
  Scaling,Week 2 | -0.11 (1.13)
  Scaling,Week 4 | -0.04 (0.74)
  Scaling,Week 8 | -0.18 (1.12)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were reported throughout the study (from Baseline Up to Week 8)
Description: Intent-to-treat analysis set was used to report adverse events.
Arm/Group | MAXCLARITY II
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAXCLARITY II (N=28)
Hiatus hernia (Gastrointestinal disorders) | 1
Application Site Burning (General disorders) | 1
Bronchitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.